CLINICAL TRIAL: NCT03458793
Title: Physical Activity Intervention for Loneliness (PAIL) in Community-dwelling Older Adults: a Feasibility Study
Brief Title: Physical Activity Intervention for Loneliness
Acronym: PAIL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Birmingham (Other)
Responsible Party: Principal Investigator, Anna Whittaker, Professor, University of Birmingham
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ERN_16-1419
Record Dates: First submitted 2018-01-23; First posted 2018-03-08 (Actual); Last update posted 2019-04-18 (Actual); Status verified 2019-04

CONDITIONS: Loneliness; Ageing; Physical Activity
Keywords: randomised controlled study; physical activity; loneliness
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: This will be a two-arm randomised controlled trial (RCT) with a wait-list control group
Who Masked: Participant
Masking Description: Computerised randomisation will be performed by an external researcher not involved in the delivery of the intervention or outcome assessment. Participants who will be assessors of their psychosocial outcomes using self-report questionnaires will be blind to the allocation concealment at the time of completing the initial questionnaires. Intervention providers who will be responsible for outcome assessments will not be blind to the intervention assignment as this would not be possible given the study and walks will be conducted by the PhD student.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The experimental group (Experimental): The experimental group will take part in the 12 week intervention after randomisation consisting of group walking and educational workshops performed once weekly for up to 90 minutes in total for each session.
  Interventions: Behavioral: Group walking and group educational workshops
- The control group (No Intervention): The control group will be a wait-listed arm that will be offered an intervention at 12 weeks after the randomisation (the delayed intervention).

INTERVENTIONS:
Behavioral: Group walking and group educational workshops — The experimental group will take part in 12 week intervention consisting of group walking and group educational workshops.
  Group walking sessions will run once weekly for up to 45 minutes each in small groups (up to 8-9 people per group) and will be delivered by a trained walk leader once weekly for duration up to 45 minutes per session.
  Group educational workshops will be delivered in the form of a group presentation once weekly for up to 45 minutes by the research team (i.e. the PhD student) on a variety of topics focused on the healthy ageing, such as eye hygiene, mental health and well-being, preventing falls, social support, nutritional guides, physical activity recommendations for older adults and other topics
  Arms: The experimental group

SUMMARY:
The purpose of this study will be to examine the feasibility of a Physical Activity Intervention for Loneliness (PAIL) in community-dwelling older adults. The research is a feasibility study designed as a two-arm randomised controlled trial (RCT) with a wait-list control group (intervention will be offered at 12 weeks to control group).

DETAILED DESCRIPTION:
After an initial screening for the eligibility based on current physical activity and levels of loneliness, up to 40 eligible participants will be randomised into the experimental or control group. Participants in the intervention group will be offered a 12-week outdoor group walking and health education workshops intervention. Each session will be performed once weekly for up to 90 minutes per session. Participants in the control group will be asked to maintain their current level of physical activity. Baseline and immediate post-intervention assessments will include anthropometry (height, weight, BMI), assessment of the resting blood pressure, physical activity for a 7-day period using accelerometer, questionnaires to assess loneliness, social support, social networks, social contacts, anxiety and depression, and expected outcomes of, and barriers to, exercise. Focus groups with participants will be conducted at 4 weeks mid-point and post-intervention to assess how the intervention might be improved; focus group transcripts will be thematically analysed using a phenomenological approach.

ELIGIBILITY:
Inclusion Criteria:

1. community-dwelling older adults aged 60 years and older as defined according to the United Nations standard numerical criterion (World Health Organization, 2016);
2. previously sedentary (i.e. engaged in less than 20 minutes per week of regular physical activity for the past month and < 125 minutes/week of moderate intensity physical activity) (Stevens et al., 1998). Moderate intensity activity that is noticeable accelerates the heart rate and is equal to approximately 3-6 metabolic equivalents (METs) (American College of Sports Medicine, 2013);
3. at risk of feeling socially isolated or lonely (indicated by a score of 6 or higher out of 9) on the 3-item loneliness scale for the phone screening by Hughes et al. (2004) (Appendix 1 - Phone-based eligibility screening form);
4. physically mobile as measured using the Short Physical Performance Battery (SPPB) (Guralnik et al., 1994) with a score ≥ 9 out of 12 (Pahor et al., 2014);
5. healthy or having one or more common chronic diseases but ambulatory;
6. without a cognitive disability as assessed by the Montreal Cognitive Assessment (MOCA) (Nasreddine et al., 2005) with a score ≥ 22 out of 30 (Freitas et al., 2013);
7. able to give written informed consent;
8. English speaking and able to complete paper and pencil questionnaires.

Exclusion Criteria:

1. not community-dwelling older adults 60 years or over;
2. not previously sedentary;
3. currently taking part in another physical activity intervention;
4. not at risk for feeling socially isolated or lonely (i.e. score of less than 6 (out of 9) on the 3-item loneliness scale for the phone screening by Hughes et al., (2004);
5. moderate to severe cognitive disability or clinical diagnosis of dementia;
6. physical disability (i.e. SPPB score less than 9);
7. severe frailty or any chronic health condition that precludes participation in the physical activity intervention and significantly limits the physical mobility of the participant (i.e. hospital settings/ non-ambulatory regime);
8. cognitive disability (i.e. less than 14 points on MOCA);
9. not able to give written informed consent;
10. not English speaking that precludes taking pen and paper tests.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2018-01-04 (Actual); Primary Completion 2018-12-28 (Actual); Study Completion 2018-12-29 (Actual)

PRIMARY OUTCOMES:
Attendance | 12 months
  Attendance will be calculated as the total number of attended sessions divided by the total number of sessions of the intervention and recorded as a percentage.
Recruitment rate | 12 months
  Percent of subjects responding to ads and friends' referrals out of total number of invitations given out as a percentage
Retention rate | 12 months
  Number of participants completing the study as a proportion of those randomised
The appropriateness and practicality of the designed intervention in the proposed settings | 12 months
  Is intervention effective for reducing loneliness, is intervention practical in the proposed design settings as assessed during the focus group interviews and analysed qualitatively
The acceptability of the intervention by participants and willingness to participate | 12 months
  Focus group interviews using phenomenological inductive approach will be aimed to help the research team to improve the quality of the delivered intervention by making changes in the methodology and design of the intervention for the future implementation in a consequent study
The assessment rate of questionnaires | 12 months
  The assessment rate of questionnaires will be evaluated as the total number of completed questionnaires divided by the total number of questionnaires and recorded as a percentage
The appropriateness of statistical methods of data analysis | 12 months
  The appropriateness of statistical methods of data analysis will be analysed by research team
Likely required sample size for the future pilot trial | 12 months
  A power calculation and sample size estimation will be calculated for meaningful outcomes (e.g. loneliness or social support) using the method based on the differences in means between the intervention and control group using the G-power software
The effect size will be calculated for loneliness | 12 months
  Means (M) and standard deviations (SD) will be used to investigate the effect size for change in loneliness using mixed between (intervention group) and within (time) repeated-measures analysis of variance (ANOVAs) with post-hoc comparisons
The effect size will be calculated for social support | 12 months
  Means (M) and standard deviations (SD) will be used to investigate the effect size for change in social support using mixed between (intervention group) and within (time) repeated-measures analysis of variance (ANOVAs) with post-hoc comparisons
The effect size will be calculated for social networks | 12 months
  Means (M) and standard deviations (SD) will be used to investigate the effect size for change in social networks using mixed between (intervention group) and within (time) repeated-measures analysis of variance (ANOVAs) with post-hoc comparisons
The effect size will be calculated for depression | 12 months
  Means (M) and standard deviations (SD) will be used to investigate the effect size for change in depression using mixed between (intervention group) and within (time) repeated-measures analysis of variance (ANOVAs) with post-hoc comparisons
The effect size will be calculated for anxiety | 12 months
  Means (M) and standard deviations (SD) will be used to investigate the effect size for change in anxiety using mixed between (intervention group) and within (time) repeated-measures analysis of variance (ANOVAs) with post-hoc comparisons
The effect size will be calculated for self-efficacy for exercise | 12 months
  Means (M) and standard deviations (SD) will be used to investigate the effect size for change in self-efficacy for exercise using mixed between (intervention group) and within (time) repeated-measures analysis of variance (ANOVAs) with post-hoc comparisons
The effect size will be calculated for satisfaction with level of social contacts | 12 months
  Means (M) and standard deviations (SD) will be used to investigate the effect size for change in satisfaction with level of social contacts using mixed between (intervention group) and within (time) repeated-measures analysis of variance (ANOVAs) with post-hoc comparisons
The effect size will be calculated for expected outcomes and barriers for exercise | 12 months
  Means (M) and standard deviations (SD) will be used to investigate the effect size for change in expected outcomes and barriers for exercise using mixed between (intervention group) and within (time) repeated-measures analysis of variance (ANOVAs) with post-hoc comparisons

SECONDARY OUTCOMES:
Loneliness | 12 months
  Loneliness will be assessed using the 8-item UCLA (University of California, Los Angeles) Loneliness Scale (UCLA-8) (Hays and DiMatteo, 1987). Items will be rated on the 4-grade Likert scale ranging from 1 (never) to 4 (often). The total scoring is ranged from a minimum of 8 to a maximum of 32 with the higher score indicating more loneliness considered to be a worse outcome. Questions "I am an outgoing person" and "I can find companionship when I want it" will be reverse scored.
Social support | 12 months
  Social support will be assessed using the 20-item Medical Outcomes Study Social Support Survey (MOSSSS) (Sherbourne and Stewart, 1991). The questionnaire will consist of 20 items including the assessment of a structural social support (number of close friends - item 1) and assessment of functional social support (items 2-20). Participants will be asked to complete the questionnaire using the five-point Likert scale ranging from low social support "None of the time" (1 point) to a high social support "All of the Time" (5 points). The total score will be calculated as the sum of the scores. Higher scores of support will show better social support.
Social networks | 12 months
  Social networks will be assessed using the 6-item Lubben's Social Network Scale (LSNS-6) (Lubben et al., 2006).LSNS-6 has total 6 items divided into two subscales: family and friendship (three items for each). The total score will be calculated by sum of the six items with scores ranging from 0 to 30. A sum of scores for six items less than 12 will indicate that the respondent had fewer than two people for social interactions. Similarly, a cut-point score of 6 on the three-item will indicate as being at risk for social isolation (Lubben et al., 2006). The family subscale will indicate that the participants had less than two family members to perform social interactions, similarly for the friendship subscale.
Depression and anxiety | 12 months
  Depression and anxiety will be assessed using the 14-item Hospital Anxiety and Depression Scale (HADS) (Zigmond and Snaith, 1983).The questionnaire consists of 14 items with the assessment on four-point scale (0-3). The maximum total score for each subscale will be 21 points. The cut-offs for the total score for each sub-scale will be: 0-7 - normal, 8-11 - mild, 12-14 - moderate, 15 and over - severe.
Self-efficacy for exercise | 12 months
  Self-efficacy for exercise will be measured using the revised 9-item Self-Efficacy for Walking/Exercise Scale (SEE) in a paper-and-pencil format (Resnick and Jenkins, 2000). Using numbers from 0 (not confident) to 10 (very confident) participants will be asked to rate their confidence in their ability to walk/exercise for 20 minutes three times per week (Resnick and Jenkins, 2000). The scoring will be calculated by summing the numerical ratings for each response and dividing by the total number of items.
Satisfaction with level of social contacts | 12 months
  Satisfaction with level of social contacts will be measured with the question "How satisfied are you with your social contacts?" (Fokkema and Knipscheer, 2007). Participants will rate their answer on a scale from 0 (entirely dissatisfied) to 10 (entirely satisfied).
Expected outcomes and barriers for exercise | 12 months
  Expected outcomes and barriers for exercise will be administered using the Expected Outcomes and Barriers for Habitual Exercise scale (Steinhardt and Dishman, 1989). Participants will be replying using the five-point Likert scale ranging from "Strongly disagree" (1 point) to "Strongly agree" (5 points). Scoring for each subscale will be provided by summing all numerical ratings for each item and divided by the total number of items. The total score of expected outcomes and barriers for exercise will be ranged from 1 point (low) to 5 points (high).
Accelerometry | 12 months
  Physical activity will be measured using ActivPAL accelerometers (PAL Technologies Ltd. Glasgow, UK). Data will be exctracted for average step counts (steps/day), time stepping (hours), time sitting/lying (hours), and energy equivalent (METs) and analysed as continuos variable for pre-to post-intervention differences.

CONTACTS AND LOCATIONS:
Overall Officials: Anna C. Whittaker, Professor, Principal Investigator — University of Birmingham
Locations (1):
- School of Sport, Exercise & Rehabilitation Sciences, University of Birmingham, Birmingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shvedko AV, Thompson JL, Greig CA, Whittaker AC. Physical Activity Intervention for Loneliness (PAIL) in community-dwelling older adults: a randomised feasibility study. Pilot Feasibility Stud. 2020 May 23;6:73. doi: 10.1186/s40814-020-00587-0. eCollection 2020. PMID 32489675
- [Derived] Shvedko AV, Thompson JL, Greig CA, Whittaker AC. Physical Activity Intervention for Loneliness (PAIL) in community-dwelling older adults: protocol for a feasibility study. Pilot Feasibility Stud. 2018 Dec 19;4:187. doi: 10.1186/s40814-018-0379-0. eCollection 2018. PMID 30598833